CLINICAL TRIAL: NCT00003877
Title: A Phase I/II Study in Metastatic Breast Cancer Patients Infused With Stromagen and Isolated, Mobilized, Autologous Peripheral Blood CD34+ Progenitor Cells After High-Dose Chemotherapy
Brief Title: Peripheral Stem Cell Transplantation With or Without Stromagen Following Chemotherapy in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Phillip McCarthy, MD, Roswell Park Cancer Institute
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067043; P30CA016056 (NIH); RPCI-DS-9828; CWRU-OSIR-1198; OSIRIS-101; NCI-G99-1516
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Paclitaxel; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: paclitaxel
Drug: thiotepa
Procedure: in vitro-treated bone marrow transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy and kill more tumor cells. It is not yet known whether Stromagen improves the success of stem cell transplantation in women with breast cancer.

PURPOSE: Randomized phase I/II trial to study the effectiveness of Stromagen during stem cell transplantation following chemotherapy in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of expanded mesenchymal stem cells (Stromagen) infusion and autologous CD34+ peripheral blood stem cells transplantation after high dose chemotherapy in women with metastatic breast cancer. II. Compare the time to neutrophil and platelet engraftment in patients receiving different doses of Stromagen. III. Evaluate the immune reconstitution of these patients after this therapy.

OUTLINE: This is a randomized, placebo controlled, blinded study. Patients are randomly assigned to one of three treatment arms. All patients undergo mobilization of peripheral blood stem cells (PBSC) using cyclophosphamide IV over 1 hour and paclitaxel IV over 3 hours on day 1, and filgrastim (G-CSF) subcutaneously beginning on day 4 and continuing until completion of leukapheresis. PBSC and bone marrow cells are collected and CD34 positive cells are then selected. About 4 weeks later, patients receive high dose chemotherapy. Cyclophosphamide IV over 24 hours, carboplatin IV over 24 hours, and thiotepa IV over 24 hours are administered on days -7 to -4. Patients then receive placebo or one of two doses of expanded mesenchymal stem cells (Stromagen) IV on day -1 and CD34+ selected PBSC IV over 2 hours on day 0. Patients are followed at 6 weeks and 12 weeks, than at 1 year.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic breast cancer involving at least 1 bone site Completed induction chemotherapy No active CNS disease Hormone receptor status: Estrogen receptor and progesterone receptor negative OR Hormone refractory disease

PATIENT CHARACTERISTICS: Age: 18 to 64 Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC greater than 1000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Hepatitis B surface antigen negative Hepatitis C negative No cirrhosis Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: Cardiac ejection fraction greater than 50% by MUGA Pulmonary: DLCO greater than 50% Other: Not pregnant Fertile patients must use effective contraception No active infection No active alcohol or substance abuse within 6 months At least 1 year since clinically significant CNS disease or seizures HIV negative No other medical condition that would preclude evaluation of the patient

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: See Disease Characteristics Radiotherapy: At least 3 years since prior radiotherapy, except local adjuvant therapy Surgery: Not specified

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-09; Primary Completion 2000-02 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Study Chair — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ireland Cancer Center, Cleveland, Ohio